CLINICAL TRIAL: NCT04548544
Title: A Randomized Controlled Feasibility Study of Emotional Well-being of Adolescents Undergoing a Mindfulness Training During the COVID-19 Pandemic
Brief Title: A Study of Adolescents Undergoing a Mindfulness Training During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-29083 (b)
Record Dates: First submitted 2020-09-11; First posted 2020-09-14 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TARA training (Experimental)
  Interventions: Behavioral: Training for Awareness, Resilience, and Action (TARA)
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Training for Awareness, Resilience, and Action (TARA) — This will be a 12-week group meditation training - Training for Awareness, Resilience, and Action (TARA)
  Arms: TARA training

SUMMARY:
The COVID-19 pandemic has been significantly affecting people's lives around the globe. Social distancing, self-quarantine, shelter-in-place measures, economic challenges, and COVID-19-cased illness and deaths have the potential to significantly impact mental health and cause stress, anxiety, and depression. Adolescents may be especially vulnerable to this situation, due to their increased vulnerability to the onset of depression and anxiety in general.

One promising approach to reduce anxiety and depression in youth is a neuroscience-based mindfulness intervention Training for Awareness Resilience and Action (TARA). TARA is usually delivered over 12 weeks by two facilitators in groups of 10-15 adolescents in-person, and it has been shown to reduce symptoms of depression and anxiety in depressed adolescents and modify brain properties. The TARA intervention can also be delivered remotely. Other types of therapy delivered remotely, such as internet-based cognitive behavioral therapy, have shown comparable efficiency to face-to-face delivery.

The objective of this study is to utilize an individually randomized group treatment, open-label, waitlist-controlled clinical trial to test the feasibility of TARA (delivered partially over Zoom) in improving the self-reported emotional well-being primary outcome (emotional problems measured with the Strengths and Difficulties Questionnaire [SDQ]) in healthy adolescents between the ages of 14 to 18 years old during the COVID-19 pandemic.

Our central hypothesis is that emotional well-being of adolescents in the intervention group will improve stronger (or deteriorate less) than in the control group. We will test this hypothesis in 21 adolescents randomized to the TARA intervention (partially delivered over Zoom) (12 adolescents) or to the waitlist control group (9 adolescents).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adolescents, 14-18 years old
* Fluency in English

Exclusion Criteria:

* Subjects younger or older than 14-18 years old.
* Subjects who are not healthy. Subjects who are taking any psychotropic medication.
* MRI contraindications (ferromagnetic objects on or inside the body, e.g., braces) and pregnancy.
* Not allowable: Current mindfulness training (e.g. MBSR, MBCT, DBT) and/or practice with a typically sitting meditation or yoga of 20 or more minutes two or more times per week within 60 days prior to study entry.
* Potential adolescent subjects with current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to the study requirements will be excluded and not allowed to enter the study.
* Potential subjects with an inability or unwillingness to give written informed assent or whose legal guardian/representative are unable or unwilling to give written informed consent will be excluded and not allowed to enter the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Tymofiyeva, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: passive control
Period: Overall Study
Arm/Group | TARA Training | Control
Started | 12 | 9
Completed | 12 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TARA Training | Control | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (1.0) | 15.7 (1.4) | 15.9 (1.2)
Sex/Gender, Customized [Count of Participants; unit: Participants] — male, female, other
  Participants
    male | 6 | 3 | 9
    female | 6 | 5 | 11
    other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 1 | 3
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21
SDQ emotional symptoms [Mean (Standard Deviation); unit: units on a scale] — The Strengths and Difficulties Questionnaire (SDQ) measures emotional and behavioral problems. Total raw scores range from 0-50. We transformed these raw SDQ scores into t-scores, a standardized score that indicates how many standard deviations a particular data point is away from the mean, which range from 0-100. Higher scores indicate more problems.
  units on a scale | 56.9 (10.0) | 57.3 (10.9) | 57.1 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in SDQ Emotional Problems
Description: Change in the level of emotional problems measured with the Strengths and Difficulties Questionnaire (SDQ). The emotional problems scores have a possible range of 0 to 100. Higher scores represent higher levels of emotional problems.
Time Frame: Baseline/randomization and 12 weeks after baseline/randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TARA Training | Control
Number analyzed (Participants) | 12 | 9
units on a scale | 2.08 (5.53) | -4.49 (4.71)
Statistical Analysis 1: Comparison: TARA Training vs Control; timepoint × group interaction; Test type: Other; p = 0.38, ANOVA; timepoint × group interaction F = 0.77, p = 0.38

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Solicited adverse events in TARA participants were captured as follows: before each TARA session participants were asked through a questionnaire: "Has there been any significant unfavorable change in your mental or physical health since last class?"; if the participant answers "yes" to this question, then the research assistant or another study staff member asked the participant for additional details regarding the participant's answer and this information was recorded in the Adverse Event form.
Arm/Group | TARA Training | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT04548544/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT04548544/ICF_001.pdf